CLINICAL TRIAL: NCT01539733
Title: Early Recognition and Optimal Treatment of Delirium in Patients With Advanced Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, H.M.W. Verheul, Prof. dr., Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009/225; 2009-013403-55 (EudraCT Number); NTR2559 (Other: Nederlands Trial Register)
Record Dates: First submitted 2012-02-21; First posted 2012-02-27 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Delirium; Advanced Cancer
MeSH Terms: conditions — Delirium | interventions — Olanzapine; Haloperidol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olanzapine (Experimental)
  Interventions: Drug: Olanzapine
- Haloperidol (Active Comparator)
  Interventions: Drug: Haloperidol

INTERVENTIONS:
Drug: Olanzapine — After randomisation to olanzapine treatment, olanzapine will be started at an initial dose of 2,5 - 5 mg orally or intramuscularly, after 2 hours subsequent titration of dosage will be based on clinical judgement with a maximum of 20 mg per 24 hours divided over a maximum of 3 gifts. Sustenance dose will consist of half of the total titrated dose per 24 hours in one gift.
  Other Names: Zyprexa
  Arms: Olanzapine
Drug: Haloperidol — After randomisation to haloperidol treatment, haloperidol dosing will be titrated, with repeated dosing of 0,5 - 2mg orally or subcutaneously every 40 minutes until signs of delirium diminish, with a maximum of 20 mg orally or 10 mg subcutaneously per 24 hours. Sustenance dose will consist of half of the total titrated dose per 24 hours in one or two gifts.
  Other Names: Haldol
  Arms: Haloperidol

SUMMARY:
The investigators designed a randomised multicenter clinical trial for patients with advanced cancer who are admitted to the medical oncology ward or high-care hospice. On admission all patients with advanced cancer will be asked to participate in this study. Consenting patients will be submitted to delirium observation screening according to the DOS. Subsequently DOS screening will be performed twice weekly until discharge. Each patient who's score is > 3 (DOS positive) is showing significant symptoms of delirium and will be submitted to the revised Delirium Rating Scale (DRS-R-98) to confirm diagnosis. To test validity of the DOS scale for this particular population, each DOS positive score will be randomly matched with a patient with a DOS score < 3 (DOSnegative) and this patient will also be submitted to DRS-R-98. When diagnosis of delirium is confirmed by DRS-98, patients will be randomised between treatment of delirium with olanzapine or haloperidol (usual care). Treatment in both groups will consist of identification and management of underlying aetiologies of delirium if possible and adding neuroleptic medication for symptom control. Patients who recover from their delirium episode as well as their caregivers will be asked to complete the Delirium Experience Questionnaire (DEQ) to assess recall of the delirium experience and the degree of distress related to the delirium episode.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with advanced cancer
* Age ≥ 18
* Patient or his / her significant other speaks Dutch fluently

Exclusion Criteria:

* Delirium is due to alcohol withdrawal
* Patient has been diagnosed with glaucoma, Parkinson's disease or dementia
* Patient is being treated with other neuroleptic medication or lithium
* Patient has another psychiatric disorder that is considered (by investigator) to interfere with assessment of delirium
* Patient had a QTc-interval of > 480 msec on ECG made on admission to the medical oncology ward (ECG is not required if patient is admitted to a high-care hospice)
* Patient has a history of neuroleptic malignant syndrome
* Patient has a history of convulsions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2010-03; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
DRS-R-98 severity rating score | Until clearance of the delirium signs or for a maximum of 2 weeks
  Primary endpoint for this trial is a DRS-R-98 severity rating score <15,25, as this is a measure for establishing clearance of delirium.

SECONDARY OUTCOMES:
Delirium resolution rate | Until clearance of the delirium signs or for a maximum of 2 weeks
  Secondary endpoint is the amount of time elapsed between start of treatment and diminishing of the signs of delirium (DOS <3, DSR-R-98 <15,25).

CONTACTS AND LOCATIONS:
Overall Officials: Henk MW Verheul, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (2):
- Netherlands (2):
  - VU University Medical Center, Amsterdam
  - Spaarne Hospital, Hoofddorp

REFERENCES:
- [Derived] van der Vorst MJDL, Neefjes ECW, Boddaert MSA, Verdegaal BATT, Beeker A, Teunissen SCC, Beekman ATF, Wilschut JA, Berkhof J, Zuurmond WWA, Verheul HMW. Olanzapine Versus Haloperidol for Treatment of Delirium in Patients with Advanced Cancer: A Phase III Randomized Clinical Trial. Oncologist. 2020 Mar;25(3):e570-e577. doi: 10.1634/theoncologist.2019-0470. Epub 2019 Dec 8. PMID 32162816
- [Derived] Neefjes ECW, van der Vorst MJDL, Boddaert MSA, Verdegaal BATT, Beeker A, Teunissen SCC, Beekman ATF, Zuurmond WWA, Berkhof J, Verheul HMW. Accuracy of the Delirium Observational Screening Scale (DOS) as a screening tool for delirium in patients with advanced cancer. BMC Cancer. 2019 Feb 19;19(1):160. doi: 10.1186/s12885-019-5351-8. PMID 30782151